CLINICAL TRIAL: NCT01638078
Title: Thalidomide fOr the Prevention of Restenosis After Coronary ArtERy Stent Implantation - The TOP RACER Trial
Brief Title: Thalidomide fOr the Prevention of Restenosis After Coronary ArtERy Stent Implantation
Acronym: TOP RACER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 429/2012/D
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary restenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide (Active Comparator): Thalidomide
  Interventions: Drug: Thalidomide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide — Thalidomide, pill, 50 mg, once p.d., 6 weeks
  Other Names: Thalidomide Celgene
  Arms: Thalidomide
Drug: Placebo — Placebo, pill, once p.d., 6 weeks
  Arms: Placebo

SUMMARY:
Percutaneous coronary intervention (PCI) with the use of bare metal stents is associated with restenosis in approximately 10% to 50% of cases.

Stenting may induce endothelial damage/dysfunction and inflammatory reactions, which in turn delay healing and endothelialization and may lead to restenosis and atherosclerosis within the stented segments.

The sedative and antinausea drug thalidomide has been shown to have both anti-inflammatory and antioncogenic properties that could be of benefit in case of PCI with stenting.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) with the use of bare metal stents is associated with restenosis in approximately 10% to 50% of cases.

Stenting may induce endothelial damage/dysfunction and inflammatory reactions, which in turn delay healing and endothelialization and may lead to restenosis and atherosclerosis within the stented segments.

Indeed, experimental studies indicate a marked activation of inflammatory cells at the site of stent struts, which is likely to play a key role in the process of neointimal proliferation and restenosis. Indeed, tumor necrosis factor and interleukins 1 and 6 are powerful stimuli for smooth muscle cell proliferation.

The sedative and antinausea drug thalidomide has been shown to have both anti-inflammatory and antioncogenic properties that could be of benefit in case of PCI with stenting.

The primary objective of this study is to carry out a double-blind, randomized, placebo-controlled study to assess the effects of oral thalidomide on restenosis rate after successful stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* A de novo native coronary artery lesions (reference vessel diameter:2.5-3.75 mm)
* Class I indication to elective percutaneous coronary intervention
* Stable conditions and no recent acute coronary syndromes
* Normal baseline values of markers of myocardial damage (creatine kinase, creatine kinase-MB, myoglobin, and troponin I)
* Able to understand and willing to sign the informed CF
* Contraindications to DES Use (Clinical history difficult to obtain, Expected poor compliance with DAPT, Non-elective surgery required, Increased risk of bleeding
* Allergy to ASA or clopidogrel/prasugrel/ticagrelor, Indication for long-term anticoagulation, Large Vessels, Focal Lesions)

Exclusion Criteria:

* Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT
* Indications to DES Use (Small Vessels, Long Lesions Diabetes, In-Stent Restenosis, Complex lesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of binary restenosis 6 months after PCI | 6 months
  6-month angiographic evidence of binary restenosis (defined as an in-stent stenosis _50% at follow-up coronary angiography)

SECONDARY OUTCOMES:
Major adverse cardiac events 6 months after PCI | 6 months
  6-month incidence of major adverse cardiac events (MACE-death, myocardial infarction, target vessel revascularization)